CLINICAL TRIAL: NCT04577157
Title: Effectiveness of mHealth Intervention Using Multifaceted Educational and Reminder Module Intervention to Improve Medication Adherence and Treatment Outcome Among Hypertensive Patients in Lahore, Pakistan: a Randomized Controlled Trial
Brief Title: mHealth App Intervention to Improve Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD, student, department of community medicine, faculty of medicine & health sciences, UPM, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DPUTRA
Record Dates: First submitted 2020-05-24; First posted 2020-10-06 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Medication Adherence; Adherence, Treatment
MeSH Terms: conditions — Medication Adherence; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: It is a parallel-design, intention-to-treat, two-arm, randomized controlled trial, six months of duration with intervention module intervention pre-test and post-test evaluations to assess the effectiveness of mHealth application using Multi-aid-package intervention(voice, written message, and multimedia picture) to improve adherence to medication in hypertensive patients in Lahore, Pakistan. Participants will be assigned to the two groups in a parallel fashion in a ratio of 1:1. The intervention group will be given a reminder module intervention and control group with standard care (as per being practiced routinely in the hospitals).
Who Masked: Investigator
Masking Description: Single-blinded The investigators will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): The participants in the intervention group will receive Health@click (seven-item multifaceted educational and reminder module) through "WhatsApp". This will be included daily notes for medication reminders, voice messages, Graphics-based Reminders (GBR), Twice-weekly Graphics-based Messages (GBM), and once-weekly lifestyle advice through video in addition to standard care (as being practiced routinely in the hospitals). Besides this, a 24/7 help provision service will be given to the participants. A qualified doctor will be there to provide this educational support. Support will be including the dose of medicine, frequency, mode of action, effects of medicine on current illness, side effects and interaction with different foods, and psychological support to the participants who feel the need.
  Interventions: Behavioral: mHealth using"WhatsApp" multifaceted educational and reminder module intervention to improve adherence
- Control Arm (No Intervention): Participants in the control group will receive no intervention except in standard care (as per being practiced routinely in the hospitals).

INTERVENTIONS:
Behavioral: mHealth using"WhatsApp" multifaceted educational and reminder module intervention to improve adherence — This multifaceted educational and reminder module is named "Health@click". The content of the reminder module has been made based on "The Health Belief Model and self-determination theory.
  1. Daily notes for medication reminders,
  2. Daily a voice message with the same content will be delivered.
  3. Daily Graphics-based Reminder (GBR).
  4. Twice-weekly Graphics-based Messages (GBM) according to Health believe model and Self-determination theory constituents.
  5. Once-weekly lifestyle advice through video
  6. Hypertension at a glance, complete information will be provided(Optional)
  7. 24/7 help provision service will be given to the participants. A qualified doctor will be there to provide this educational support. Support will be including the dose of medicine, frequency, mode of action, effects of medicine on current illness, side effects, and interaction with different foods (Optional).
  Other Names: Mobile health intervention, reminder module intervention,
  Arms: Intervention Arm

SUMMARY:
It is a parallel-design, two-arm, randomized controlled trial designed to assess the effectiveness of mHealth application using 7- items, multifaceted educational and reminder module intervention( written message, voice message, multimedia picture, Graphic based Messages(GBM), video, hypertension at a glance, and doctor support) to improve adherence to medication in hypertensive patients and clinical outcome systolic blood pressure in Lahore, Pakistan. Cost-effectiveness of this study will also be done.

DETAILED DESCRIPTION:
Hypertension is indeed a significant public health concern in Pakistan. Hypertension drastically affects 18.9% of adolescents of age greater than 15 and 33% of adults of age above 45. Uncontrolled blood pressure (BP) is a leading risk factor for major hypertensive complications. In Pakistan, suboptimal adherence to medication remains a stumbling block to the success of antihypertensive treatment. A majority of the population in Pakistan on treatment is found to be non-adherent. mHealth is quite an apt tool positioned to counter these challenges of poor adherence in resource limit settings like Pakistan. What is available is too little to establish any causal relationship. The aim of this study is to assess the effectiveness of mHealth intervention by using a reminder module in improving patient medication adherence in hypertensive patients. The intervention was designed to improve the hypertension-related adherence in participants in the intervention group. The module will be developed and undergone via the process of consultations from a group of experts. These will include professors of epidemiology, one expert in behavioral intervention, two professors of health education, and one cardiologist specialist in hypertension management. For the intervention group, a "multifaceted educational reminder module" will be developed and delivered through "WhatsApp" (written message, voice message, and Graphic-based Reminder (GBR)) by an Information and Technology (IT) facilitator. This will be included daily notes for medication reminders, voice messages,s and Graphic-based Reminders (GBR), Twice-weekly Graphic based Messages(GBM), Lifestyle changing video, hypertension at a glance, and doctor support in addition to the standard care (as per being practiced routinely in the hospitals). WhatsApp is used in this study because of its feature of ticks, which turns out to blue after seeing the message and it is an indication to the sender if the receiver has seen the message, so, the participants no longer need to respond to calls or messages. If the intervention is found effective, it can help in developing educational guidelines for patients to improve their medication adherence and reduce related complications at the same time. This study will give a new line of research for coming researchers in the long run. Moreover, its cost-effectiveness will be assessed to predict one dollar bring about improvement per mmHg.

ELIGIBILITY:
Inclusion criteria

* Participants with age more than 18 years
* Patients diagnosed with essential hypertension and registered in the cardiology and medical Outpatient Departments (OPDs) of three tertiary care hospitals of Lahore for the last one month.
* Participants on antihypertensive medication
* Only one member from one family.
* Participants have a mobile phone and have "Whatsapp" application installed on their cell phones
* Participants who can operate a mobile phone and can read and send a message on "Whatsapp".

Exclusion Criteria

* Participants with planned travel within two months with no mobile signals.
* Participants with a history of malignancy and require medication adjustment.
* Participants with any planned procedure (during the study period) demand immediate medication changes like CABG, PCI, or CEA (Carotid Endarterectomy)
* Participants who are suffering from dementia, depression (self-reporting)
* Participants with blood-pressure measurement of >220/>120 mmHg (symptoms of a hypertensive emergency)
* Participants who are pregnant (self-reporting)
* Participants who are in their lactation period
* Participants within 3 months postpartum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Adherence to medication (Medication Adherence Score)- Self Reported Scale | 6- month from baseline
  The primary outcome is (change) medication adherence to antihypertensive treatment (AHT) at 6 months. This will be assessed by self-reporting using a Standardized questionnaire, Self-efficacy for Appropriate Medication Adherence Scale (SEAMS) at 0, 3, and 6 months. It is a 13-item scale with a three-point response questionnaire, with (1 _ not confident, 2 _ somewhat confident and 3 _ very confident). The potential score for the 13-item scale ranged from 13 to 39. Higher scores indicated higher levels of self-efficacy for medication adherence and vice versa. Besides SEAMS, adherence rates will be also be calculated by 'pills taken over a specific period of time, divided by pills prescribed for that specific period of time. The cut-off value of 80% is set. Less than 80% will be considered non-adherent while >80% will be adherent. It will be self-reporting.
Change in systolic blood pressure | 6- month from baseline
  The secondary outcome is a change in systolic blood pressure (SBP) of participants at 6 months. This will be assessed on measuring blood pressure at the hospital by a blinded staff nurse at 0, 3, and 6 months at the hospital by a blinded staff nurse using the calibrated upper-arm electronic sphygmomanometer (OMRON HEM-7200, OMRON Corporation, Dalian) with standard guidelines.

OTHER OUTCOMES:
Expected Outcomes | 6-months
  1. A significant difference in treatment adherence is expected in the intervention group compared to the control group. [ Time Frame: At 6-months ]
  2. Self-reported adherence to antihypertensive treatment [ Time Frame: At 6-months ]
  3. The proportion of participants with a systolic blood pressure < 140 mmHg and a diastolic blood pressure <90 mmHg [ Time Frame: At 6-months ]

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Kiran, MBBS, Study Director — Doctors Hospital, Lahore; Arshed Muhammad, MBBS, Principal Investigator — UPM
Locations (1):
- Sheikh Zayed, Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamal AK, Khalid W, Muqeet A, Jamil A, Farhat K, Gillani SRA, Zulfiqar M, Saif M, Muhammad AA, Zaidi F, Mustafa M, Gowani A, Sharif S, Bokhari SS, Tai J, Rahman N, Sultan FAT, Sayani S, Virani SS. Making prescriptions "talk" to stroke and heart attack survivors to improve adherence: Results of a randomized clinical trial (The Talking Rx Study). PLoS One. 2018 Dec 20;13(12):e0197671. doi: 10.1371/journal.pone.0197671. eCollection 2018. PMID 30571697
- [Background] Bobrow K, Farmer AJ, Springer D, Shanyinde M, Yu LM, Brennan T, Rayner B, Namane M, Steyn K, Tarassenko L, Levitt N. Mobile Phone Text Messages to Support Treatment Adherence in Adults With High Blood Pressure (SMS-Text Adherence Support [StAR]): A Single-Blind, Randomized Trial. Circulation. 2016 Feb 9;133(6):592-600. doi: 10.1161/CIRCULATIONAHA.115.017530. Epub 2016 Jan 14. PMID 26769742
- [Background] Fang R, Li X. Electronic messaging support service programs improve adherence to lipid-lowering therapy among outpatients with coronary artery disease: an exploratory randomised control study. J Clin Nurs. 2016 Mar;25(5-6):664-71. doi: 10.1111/jocn.12988. Epub 2015 Nov 1. PMID 26522838
- [Background] Kamal AK, Shaikh Q, Pasha O, Azam I, Islam M, Memon AA, Rehman H, Akram MA, Affan M, Nazir S, Aziz S, Jan M, Andani A, Muqeet A, Ahmed B, Khoja S. A randomized controlled behavioral intervention trial to improve medication adherence in adult stroke patients with prescription tailored Short Messaging Service (SMS)-SMS4Stroke study. BMC Neurol. 2015 Oct 21;15:212. doi: 10.1186/s12883-015-0471-5. PMID 26486857
- [Background] Park LG, Howie-Esquivel J, Chung ML, Dracup K. A text messaging intervention to promote medication adherence for patients with coronary heart disease: a randomized controlled trial. Patient Educ Couns. 2014 Feb;94(2):261-8. doi: 10.1016/j.pec.2013.10.027. Epub 2013 Nov 18. PMID 24321403
- [Background] Vollmer WM, Owen-Smith AA, Tom JO, Laws R, Ditmer DG, Smith DH, Waterbury AC, Schneider JL, Yonehara CH, Williams A, Vupputuri S, Rand CS. Improving adherence to cardiovascular disease medications with information technology. Am J Manag Care. 2014 Nov;20(11 Spec No. 17):SP502-10. PMID 25811824
- [Background] Wald DS, Bestwick JP, Raiman L, Brendell R, Wald NJ. Randomised trial of text messaging on adherence to cardiovascular preventive treatment (INTERACT trial). PLoS One. 2014 Dec 5;9(12):e114268. doi: 10.1371/journal.pone.0114268. eCollection 2014. PMID 25479285
- [Background] WHO | The Declaration of Helsinki and public health. (n.d.). WHO; World Health Organization. Retrieved April 11, 2020, from https://www.who.int/bulletin/volumes/86/8/08-050955/en
- [Background] Ni Z, Liu C, Wu B, Yang Q, Douglas C, Shaw RJ. An mHealth intervention to improve medication adherence among patients with coronary heart disease in China: Development of an intervention. Int J Nurs Sci. 2018 Sep 8;5(4):322-330. doi: 10.1016/j.ijnss.2018.09.003. eCollection 2018 Oct 10. PMID 31406843
- [Background] Gandapur Y, Kianoush S, Kelli HM, Misra S, Urrea B, Blaha MJ, Graham G, Marvel FA, Martin SS. The role of mHealth for improving medication adherence in patients with cardiovascular disease: a systematic review. Eur Heart J Qual Care Clin Outcomes. 2016 Oct 1;2(4):237-244. doi: 10.1093/ehjqcco/qcw018. PMID 29474713
- [Background] Jafar TH, Jafary FH, Jessani S, Chaturvedi N. Heart disease epidemic in Pakistan: women and men at equal risk. Am Heart J. 2005 Aug;150(2):221-6. doi: 10.1016/j.ahj.2004.09.025. PMID 16086922
- [Background] Lim CY, In J. Randomization in clinical studies. Korean J Anesthesiol. 2019 Jun;72(3):221-232. doi: 10.4097/kja.19049. Epub 2019 Apr 1. PMID 30929415
- [Background] Noordzij M, Tripepi G, Dekker FW, Zoccali C, Tanck MW, Jager KJ. Sample size calculations: basic principles and common pitfalls. Nephrol Dial Transplant. 2010 May;25(5):1388-93. doi: 10.1093/ndt/gfp732. Epub 2010 Jan 12. PMID 20067907
- [Background] Pednekar PP, Agh T, Malmenas M, Raval AD, Bennett BM, Borah BJ, Hutchins DS, Manias E, Williams AF, Hiligsmann M, Turcu-Stiolica A, Zeber JE, Abrahamyan L, Bunz TJ, Peterson AM. Methods for Measuring Multiple Medication Adherence: A Systematic Review-Report of the ISPOR Medication Adherence and Persistence Special Interest Group. Value Health. 2019 Feb;22(2):139-156. doi: 10.1016/j.jval.2018.08.006. Epub 2018 Oct 25. PMID 30711058
- [Background] Roberts C, Torgerson D. Randomisation methods in controlled trials. BMJ. 1998 Nov 7;317(7168):1301. doi: 10.1136/bmj.317.7168.1301. No abstract available. PMID 9804722
- [Background] Altman DG, Schulz KF. Statistics notes: Concealing treatment allocation in randomised trials. BMJ. 2001 Aug 25;323(7310):446-7. doi: 10.1136/bmj.323.7310.446. No abstract available. PMID 11520850
- [Background] Bhide A, Shah PS, Acharya G. A simplified guide to randomized controlled trials. Acta Obstet Gynecol Scand. 2018 Apr;97(4):380-387. doi: 10.1111/aogs.13309. Epub 2018 Feb 27. PMID 29377058
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Derived] Arshed M, Mahmud A, Minhat HS, Lim PY, Zakar R. Effectiveness of a Multifaceted Mobile Health Intervention (Multi-Aid-Package) in Medication Adherence and Treatment Outcomes Among Patients With Hypertension in a Low- to Middle-Income Country: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2024 Jun 19;12:e50248. doi: 10.2196/50248. PMID 38896837